CLINICAL TRIAL: NCT06553391
Title: Heart Rhythm Changes in Patients With Atrial Fibrillation After Cardiopulmonary Bypass: a Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Chen Linlin, Clinical Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: SP2023036（01）
Record Dates: First submitted 2024-07-12; First posted 2024-08-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pharmacological cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Aminophylline; Ephedrine; Isoproterenol; Amiodarone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TMR group: The treatment regimen for the tetralogy of medication regimen group (TMR group）commences with the administration of amiodarone during rewarming. In the event of cardiac relapse, a combination of the following drugs may be utilized: aminophylline, ephedrine, and isoproterenol. The selection of these medications is contingent upon the patient's blood pressure and heart rate.
  Interventions: Drug: The tetralogy of medication regimen
- Control group: Patients in the control group did not receive treatment with antiarrhythmic drugs.

INTERVENTIONS:
Drug: The tetralogy of medication regimen — During the rewarming process, the study group received an injection of 0.15g amiodarone via the extracorporeal circulation oxygenator. After heart re-beating：
  1. If the heart rate is ≥70 beats per minute without specific therapy and in sinus rhythm or atrioventricular junctional rhythm, no special treatment is required. If the heart rate <70 beats/min, intravenous injection of isoproterenol 2 ug may be administered.
  2. In cases where there is sinus rhythm or atrioventricular junctional rhythm with a heart rate <70 beats/min and perfusion pressure <60mmHg, intravenous injection of ephedrine 10 mg + aminophylline 0.15 g should be given.
  3. For patients with atrioventricular junctional rhythm or sinus rhythm and a heart rate <70 beats/min but perfusion pressure ≥60mmHg, intravenous injections of aminophylline (0.15g) and ephedrine (10 mg) .
  4. In cases where there is atrial fibrillation (AF), and the heart rate is ≥70 beats/min without special treatment.
  Other Names: aminophylline; ephedrine; isoproterenol; amiodarone
  Groups: TMR group

SUMMARY:
The goal of this observational study is to learn about the lthe effect of the tetralogy of medication regimen on intraoperative cardioversion in patients with persistent AF. The main question it aims to answer is:

Does the regimen improve the success rate of cardioversion in patients with persistent AF during cardiac surgery? The treatment protocol commences with the administration of amiodarone, followed by the administration of either all or a portion of the subsequent medications: aminophylline, ephedrine, and isoproterenol.

This observational cohort study was conducted at the Chinese Academy of Medical Sciences Fuwai Shenzhen Hospital using the electronic medical record database, from August 1, 2024, to January 1, 2025. Patients diagnosed with atrial fibrillation who underwent cardiac surgery between June 1, 2020, and December 31, 2024, were included in the study.

DETAILED DESCRIPTION:
Background: Most patients with atrial fibrillation (AF) continue to experience AF following cardiac surgery, which is not conducive to postoperative circulatory stability. Intraoperative active cardioversion has rarely studied due to uncertainty regarding the efficacy of pharmacological cardioversion and the recurrence rate of AF in patients with persistent AF.

Objective: To assess the effect of the tetralogy of medication regimen on intraoperative cardioversion in patients with persistent AF.

Methods: This observational cohort study was conducted at the Chinese Academy of Medical Sciences Fuwai Shenzhen Hospital using the electronic medical record database, from August 1, 2024, to January 1, 2025. Patients diagnosed with AF who underwent cardiac surgery between June 1, 2020, and December 31, 2024, were included in the study. These patients undergoing pharmacological cardioversion during surgery were matched with untreated patients in a 1:1 ratio based on age, sex, weight, diagnosis, beta blocker and digoxin usage, indicators from cardiac ultrasound and blood gas analysis. The treatment protocol commences with the administration of amiodarone, followed by the administration of either all or a portion of the subsequent medications: aminophylline, ephedrine, and isoproterenol. The choice between these drugs depends on the patient's blood pressure and heart rate. The incidence of cardioversion in patients who underwent the tetralogy of medication regimen approach was compared with that of untreated patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅱ-Ⅲ,
* Aged 18-70 years,
* Who were scheduled for elective cardiac surgery under general anesthesia,
* Who were diagnosed with atrial fibrillation by preoperative 12-lead electrocardiogram or 24-hour holter electrocardiogram.

Exclusion Criteria:

* Allergic to iodine, amiodarone or its excipients
* Pulmonary fibrosis
* Keratopathy or severe loss of vision or blindness
* Patients with sick sinus syndrome, severe bradycardia (heart rate <50bpm), second- or higher-degree atrioventricular block
* Preoperative intravenous infusion of amiodarone
* Intraoperative radiofrequency ablation of atrial fibrillation
* The patient is participating in another interventional clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with atrial fibrillationwho were scheduled for elective cardiac surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Sinus rhythm | From the release of the aortic cross-clamp until 12 hours after surgery
  Electrocardiogram monitoring

SECONDARY OUTCOMES:
Mean arterial pressure | From the release of the aortic cross-clamp until the end of surgery
  Invasive arterial blood pressure test
the use of temporary pacemakers | From the release of the aortic cross-clamp until 12 hours after surgery
  Postoperative record

CONTACTS AND LOCATIONS:
Overall Officials: linlin chen, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The analytical data from this study was shared upon the completion of the research. Individuals who wish to access the data are required to declare their intended use for it. Contact information for the person responsible for managing the data can be obtained from the ClinicalTrials.gov PRS website.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be made available after the study, with no deadline.
Access Criteria: Visitors must obtain permission from the study leader and declare the purpose of their data.

REFERENCES:
- [Background] Noubiap JJ, Bigna JJ, Agbor VN, Mbanga C, Ndoadoumgue AL, Nkeck JR, Kamguia A, Nyaga UF, Ntusi NAB. Meta-analysis of Atrial Fibrillation in Patients With Various Cardiomyopathies. Am J Cardiol. 2019 Jul 15;124(2):262-269. doi: 10.1016/j.amjcard.2019.04.028. Epub 2019 Apr 24. PMID 31109634
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Tarantini G, Mojoli M, Windecker S, Wendler O, Lefevre T, Saia F, Walther T, Rubino P, Bartorelli AL, Napodano M, D'Onofrio A, Gerosa G, Iliceto S, Vahanian A. Prevalence and Impact of Atrial Fibrillation in Patients With Severe Aortic Stenosis Undergoing Transcatheter Aortic Valve Replacement: An Analysis From the SOURCE XT Prospective Multicenter Registry. JACC Cardiovasc Interv. 2016 May 9;9(9):937-46. doi: 10.1016/j.jcin.2016.01.037. Epub 2016 Apr 13. PMID 27085579
- [Background] Weng LC, Preis SR, Hulme OL, Larson MG, Choi SH, Wang B, Trinquart L, McManus DD, Staerk L, Lin H, Lunetta KL, Ellinor PT, Benjamin EJ, Lubitz SA. Genetic Predisposition, Clinical Risk Factor Burden, and Lifetime Risk of Atrial Fibrillation. Circulation. 2018 Mar 6;137(10):1027-1038. doi: 10.1161/CIRCULATIONAHA.117.031431. Epub 2017 Nov 12. PMID 29129827
- [Background] Santhanakrishnan R, Wang N, Larson MG, Magnani JW, McManus DD, Lubitz SA, Ellinor PT, Cheng S, Vasan RS, Lee DS, Wang TJ, Levy D, Benjamin EJ, Ho JE. Atrial Fibrillation Begets Heart Failure and Vice Versa: Temporal Associations and Differences in Preserved Versus Reduced Ejection Fraction. Circulation. 2016 Feb 2;133(5):484-92. doi: 10.1161/CIRCULATIONAHA.115.018614. Epub 2016 Jan 8. PMID 26746177
- [Background] Kamal F, Abd Al Jawad MN, Gamal M. Efficacy of Intraoperative Low Dose Intravenous Amiodarone in Pharmacologic Cardioversion in Patients with Preoperative Atrial Fibrillation Presenting for Mitral Valve Replacement Surgery Randomized Control Trial. Heart Surg Forum. 2022 Jul 27;25(4):E564-E570. doi: 10.1532/hsf.4901. PMID 36052897